CLINICAL TRIAL: NCT03588208
Title: Evaluation of the Effectiveness of a Progressive Resistance Training Program for Patients With Fibromyalgia: a Randomized Controlled Trial
Brief Title: Progressive Resistance Training for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Anamaria Jones, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP UNIFESP 482056
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pain; Function; Quality of life
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Progressive resistance training program; Other: Educational Program
- Control Group (Active Comparator)
  Interventions: Other: Educational Program

INTERVENTIONS:
Other: Progressive resistance training program — Progressive resistance training program were performed twice a week for 12 weeks. The charge intensity was progressively increased from 40% to 80% of 1 repetition maximum. The following muscle groups were worked: trunk flexors and extensors, elbow flexors and extensors, knee flexors and extensors, hip abductors and adductors and shoulder abductors. In addition to strength training.
  Arms: Intervention Group
Other: Educational Program — Structured education program were performed during one hour class once a week for five weeks

SUMMARY:
Patients in the experimental group underwent a progressive resistance training program, performed twice a week for 12 weeks. The charge intensity was progressively increased from 40% to 80% of 1 repetition maximum. The following muscle groups were worked: trunk flexors and extensors, elbow flexors and extensors, knee flexors and extensors, hip abductors and adductors and shoulder abductors. In addition to strength training, the experimental group also conducted a structured education program in one hour class once a week for five weeks. Patients in the control group performed the same education program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia according to the criteria of the American College of Rheumatology;
* Feminine gender;
* Age between 18 and 65 years;
* Pain between 3 and 8 cm in the Numerical Pain Scale (END);
* Have not changed treatment for fibromyalgia in the past three months;
* Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Cognitive deficit that does not allow the understanding of the evaluation instruments;
* Other diseases that make it impossible to perform the exercises;
* Physical activity started or changed in the last three months;
* Physical therapy in the last six months;
* In litigation.

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-09-02 (Actual); Study Completion 2018-03-25 (Actual)

PRIMARY OUTCOMES:
Change in pain | Baseline and after 6 and 12 weeks
  Measured by numerical pain scale

SECONDARY OUTCOMES:
Change in Health related quality of life | Baseline and after 6 and 12 weeks
  Measured by Fibromyalgia Impact Questionnaire
Change in Generic quality of life | Baseline and after 6 and 12 weeks
  Measured by the Medical Outcome Survey Short Form 36
Change in Functional capacity | Baseline and after 6 and 12 weeks
  Measured by the 6-minute Walk Test
Change in strength | Baseline and after 6 and 12 weeks
  Measured by the 1 repetition maximum